CLINICAL TRIAL: NCT02759419
Title: An Open-label, Multi-national, Multi-center, Single-arm, Uncontrolled, Long-term Extension Study of Orally Administered Riociguat in Patients With Symptomatic Pulmonary Arterial Hypertension (PAH) Who Received Riociguat in a Bayer Clinical Trial
Brief Title: A Long-term Extension Study of Riociguat in Patients With Symptomatic Pulmonary Arterial Hypertension.
Acronym: RIALTO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18694; 2016-000501-36 (EudraCT Number)
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAY63-2521 (Experimental): Single-arm, uncontrolled
  Interventions: Drug: Adempas (Riociguat, BAY63-2521)

INTERVENTIONS:
Drug: Adempas (Riociguat, BAY63-2521) — 0.5 to 2.5 mg in 0.5 mg increments (according to individual adapted optimal dose determined in originating study) administered three times daily (tid)

SUMMARY:
To provide riociguat therapy to eligible patients with PAH originating from Bayer-sponsored trials with BAY63-2521/ Riociguat / Adempas® who are currently or recently treated in these trials until lack of patient benefit as assessed by investigator, or commercial availability and reimbursement.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Pulmonary Arterial Hypertension (PAH) participating or having participated in the Bayer-sponsored studies 12935, 16719 or 18588, who have completed the main study phase and are still being treated with riociguat (either while still being on treatment with the respective study drug or by commercial means with Adempas) and who, in the opinion of the investigator, are expected to continue to have an overall positive benefit/risk from continuing treatment.
* Women and men of reproductive potential must agree to use adequate contraception when sexually active. This applies for the time period between signing of the informed consent form and 30 days after the last administration of study drug.

Exclusion Criteria:

* Ongoing serious adverse event (SAE) from originating study that is assessed as related to riociguat
* Pregnant women or breast-feeding women
* Any contra-indication to Adempas treatment listed in the BAY63-2521 / Riociguat Investigators's Brochure
* Concomitant participation in another clinical study with the study drug
* Patients with pulmonary hypertension associated with idiopathic interstitial pneumonia (PH-IIP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-emergent adverse events (TEAEs) as measure of safety and tolerability | Up to approx. 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- France (5):
  - Besançon
  - Brest
  - Le Kremlin-Bicêtre
  - Lille
  - Rouen
- South Korea (2):
  - Seoul, Seoul Teugbyeolsi
  - Seoul

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — http://clinicaltrials.bayer.com/study/18694